CLINICAL TRIAL: NCT02354768
Title: Evaluation of Lanreotide Efficacity in High Output Stoma: a Multicentric Randomized Study
Acronym: ILEHOS
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Collaborators: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5971
Record Dates: First submitted 2015-01-26; First posted 2015-02-03 (Estimated); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: High Output Stoma
MeSH Terms: interventions — Smectite; Loperamide; Single Person

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lanreotide and anti-diarrheal treatments (Experimental): * Lanreotide: 1 single injection at day 0 (lanreotide 120 mg)
  * Diosmectite (3 g) 6 / day for 72 hours (fromD0 to D3)
  * Chlorhydrate of Loperamide (2 mg capsule or tablet) 6 / day for 72 hours (D0 to D3)
  * hydration
  Interventions: Drug: Effects of lanreotide with current anti-diarrheal treatments (diosmectite and loperamide)
- Current anti-diarrheal treatments alone (Active Comparator): * Diosmectite (3 g) 6 / day for 72 hours (fromD0 to D3)
  * Chlorhydrate of Loperamide (2 mg capsule or tablet) 6 / day for 72 hours (D0 to D3)
  * Hydration
  Interventions: Drug: Effects of current anti-diarrheal treatments (diosmectite and loperamide) alone

INTERVENTIONS:
Drug: Effects of lanreotide with current anti-diarrheal treatments (diosmectite and loperamide)
  Arms: lanreotide and anti-diarrheal treatments
Drug: Effects of current anti-diarrheal treatments (diosmectite and loperamide) alone
  Arms: Current anti-diarrheal treatments alone

SUMMARY:
Dehydration is a major problem of high output stoma with a 17% rate of readmission at 30 days. Dehydratations are resulting of significant electrolyte loss: sodium, potassium and renal failure. Nowadays, there are no recommendations nor national nor international for high output ileostomy treatment. Apart from the anti-diarrhea treatments used in current practice, somatostatin analogs have proven efficacy in the literature. Theses analogs permit to decrease significantly gastrointestinal secretions. Several teams use these analogs in order to decrease the flow of highly productive ileostomy.

The aim of the study is to evaluate the efficacy first line treatment with lanreotide associated with current anti-diarrheal treatment for patients with high output ileostomy (or greater throughput 1.5l / 24h) with or without associated dehydration

ELIGIBILITY:
Inclusion Criteria:

* Legal at the time of signing the agreement
* Subject affiliated to the french social protection
* Ileostomy has achieved since 10 days minimum at day 0 (D0: start of study treatment)
* Ileostomy output > 1.5 liters / 24h for at least 24 hours at day 0
* accept to use an effective method of contraception during the study: (during the 6 months following injection of lanreotide for the experimental group and for the control group: 4 days after the last dose of chlorhydrate of loperamide
* People able to understand the objectives, modalities and risks related to the study and give written informed consent

Exclusion Criteria:

* people with guardianship or with judicial protection
* simultaneous participation in another biomedical research protocol involving a drug or topic exclusion period
* pregnancy or breastfeeding
* administration of lanreotide or related peptide between surgery and D0
* hypersensitivities to lanreotide or related peptides and / or diosmectite and / or loperamide and / or one of their excipients
* acute hemorrhagic colitis
* bloody diarrhea and / or high fever
* Clostridium Difficile Infection at the inclusion
* uncontrolled diabetis defined by HbA1c> 7% at D0

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2015-10-22 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-01-26 (Actual)

PRIMARY OUTCOMES:
Number of ileostomy bags used per day | 72 hours

SECONDARY OUTCOMES:
Number of ileostomy bags used per day | from Day 0 to Day 6
Blood urea and creatinine rates | every 2 days until Day6 (Day 0, Day 2, Day 4, Day 6)
Length of stay | duration of hospital stay, an expected average of 6 days
Serious adverse events | Day 0, Day 1 Day 2, Day3, Day 4, Day 5, Day 6, 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Benoit ROMAIN, MD, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (6):
- France (6):
  - Hôpital Jean Minjoz - Service de Chirurgie Digestive, Besançon
  - Hôpitaux Civils de Colmar - Service de Chirurgie Digestive, Colmar
  - Hopital du Bocage - CHU Dijon- Service de Chirurgie Digestive, Dijon
  - Hôpital Emile MULLER - Service de Chirurgie Digestive, Mulhouse
  - CHU Robert Debré Service de chirurgie générale, digestive et endocrinienne, Reims
  - Hôpital de Hautepierre-Service de Chirurgie Digestive, Strasbourg

IPD SHARING:
Plan to Share IPD: No